CLINICAL TRIAL: NCT00894231
Title: Levocetirizine Effect on Nasal Nitric Oxide and Nasal Eosinophils in Subjects With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AAADRS Clinical Research Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Miguel J Lanz MD FAAAAI, AAADRS
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIS071108
Record Dates: First submitted 2009-04-17; First posted 2009-05-06 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Sugar tablet
  Interventions: Drug: placebo
- Xyzal (Active Comparator)
  Interventions: Drug: levocetirizine (Xyzal)

INTERVENTIONS:
Drug: levocetirizine (Xyzal) — 5mg po QD
  Other Names: Xyzal
  Arms: Xyzal
Drug: placebo — sugar tablet
  Arms: placebo

SUMMARY:
The purpose of this study is to noninvasively measure the anti-inflammatory effect of levocetirizine after two weeks of treatment in allergic rhinitis subjects.

ELIGIBILITY:
Inclusion Criteria:

* ICF signed
* Diagnosis of PAR for 6-12 months greater
* 12 years and older
* Decreased nasal NO values at baseline
* Compliance and ability to perform maneuvers and responsibilities

Exclusion Criteria:

* Oral or systemic steroids for 60 days prior
* Inhaled, nasal, nebulized steroids w/i 4 weeks
* Hospitalization or life threatening asthma
* Use of nasal or oral antihistamines w/i 4 weeks
* Upper or lower airways infection
* Direct cigarette smoke exposure

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The change in objective measure of inflammation nasal NO after LC treatment. | two weeks

SECONDARY OUTCOMES:
The change in nasal eosinophils, QOL and diary scores after LC treatment. | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miguel J Lanz, MD, Principal Investigator — AAADRS Clinical Research Center
Locations (1):
- AAADRS, Coral Gables, Florida, United States